CLINICAL TRIAL: NCT00055991
Title: A Multicenter Randomized Double-Blind Trial Of Targretin Capsules Modifying Immunophenotypic Markers Related To Breast Cancer Progression In Breast Tissue From Genetically Identified High Risk Patients
Brief Title: Bexarotene in Preventing Breast Cancer in Women at Genetic Risk
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor Breast Care Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000271913; 5U19CA086809 (NIH); NCT00206479 (obsolete NCT alias)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bexarotene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bexarotene (Experimental): Bexarotene / Targretin
  Interventions: Drug: bexarotene
- Sugar Pill (Placebo Comparator): Sugar pill / placebo
  Interventions: Drug: bexarotene

INTERVENTIONS:
Drug: bexarotene — This drug is a retinoid. The anti-tumor action of retinoids, as well as their potential in chemoprevention, supports the need to further identify the spectrum of responsive tumors, to identify the molecular mechanisms associated with retinoid action, and to identify and develop new retinoids that have unique properties and an improved therapeutic index.
  Other Names: Targretin

SUMMARY:
RATIONALE: Chemoprevention therapy uses certain drugs to try to prevent the development or recurrence of cancer. It is not yet known whether bexarotene is effective in preventing breast cancer.

PURPOSE: Randomized clinical trial to study the effectiveness of bexarotene in preventing breast cancer in women who are at genetic risk of developing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether bexarotene can modify immunophenotypic markers related to breast cancer progression in women at high genetic risk for breast cancer.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to menopausal status (women with a uterus who have not had a menstrual period for more than 1 year vs any woman over 55 years old vs women 55 years and under without a uterus whose follicle-stimulating hormone is in the postmenopausal range). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral bexarotene once daily on days 1-28.
* Arm II: Patients receive oral placebo as in arm I. In both arms, treatment continues in the absence of unacceptable toxicity or elevation of triglycerides to greater than 800 mg/dL. Patients undergo 2 breast biopsies in the same location on days 1 and 29.

Patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Known carrier of a BRCA-1 or BRCA-2 mutation

  * Copy of laboratory report stating results must be available for review OR
* At risk for carrying a BRCA-1 or BRCA-2 mutation

  * At least 10% risk by Parmigiana probability model
* Must have at least 1 breast that has never been involved with cancer and has not been irradiated
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hematocrit greater than 30%

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 1.5 times ULN
* Albumin no greater than 1.5 times ULN
* No biliary tract disease

Renal

* Creatinine no greater than 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 1 month before, during, and for 1 month after study therapy
* Triglycerides normal
* Thyroid-stimulating hormone and thyroxine normal
* Willing to undergo 2 duplicate needle biopsies of the breast
* Willing to undergo genetic testing for BRCA-1 and BRCA-2
* No uncontrolled hyperlipidemia
* No nontoxic goiter or thyroid enlargement
* No severe underlying chronic illness or disease
* No uncontrolled diabetes
* No history of pancreatitis
* No cancer within the past year except skin cancer or carcinoma in situ of the cervix (defined from the date of first diagnosis)
* No concurrent alcohol use (greater than 3 drinks or its equivalent per day)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 1 year since prior chemotherapy for a neoplasm

Endocrine therapy

* More than 3 months since prior postmenopausal hormonal therapy (including estrogens or progestins)
* More than 3 months since prior tamoxifen or other selective estrogen-receptor modulators
* No concurrent hormone replacement therapy
* Concurrent thyroid hormone supplementation allowed

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* More than 30 days since prior investigational medications
* More than 3 months since prior oral vitamin A supplements greater than the recommended daily requirement (5,000 IU) or therapeutic oral or topical vitamin A derivatives (e.g., isotretinoin)
* No concurrent participation in a study of an investigational agent
* No concurrent medications known to be associated with pancreatic toxicity or to increase triglyceride levels

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2001-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Chemopreventive effect as determine by a modification of the immunophenotypic characteristics of normal breast tissue at day 29 during study treatment and day 30 after study completion

SECONDARY OUTCOMES:
Apoptosis at day 29 during study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Elledge, MD, Study Chair — Baylor College of Medicine
Locations (4):
- United States (4):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas